CLINICAL TRIAL: NCT05759286
Title: Effect of Aromatherapy Using Lavender- Neroli Oils Blend and Music in the Management of Dental Anxiety in Children
Brief Title: A Blend of Lavender-neroli Oils Aromatherapy and Music for Managing Anxiety in a Pediatric Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Pedo-01-2023
Record Dates: First submitted 2023-02-08; First posted 2023-03-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dental Anxiety
Keywords: aromatherapy; music; lavender; neroli; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Aromatherapy; Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- aromatherapy group (Experimental): Children in this group will receive IANB injection with a nasal mask (similar to a nitrous oxide mask), the way the mask work is by putting on its circular hole a 3d printed perforated box containing cotton balls loaded with lavender-neroli oils blend
  Interventions: Behavioral: Aromatherapy
- music group (Experimental): children in this group will receive IANB injections by listening to music as background from a recorder.
  Interventions: Behavioral: Music
- combination group music and aromatherapy (Experimental): children in this group will receive aromatherapy using the nasal mask with an aromatherapy box as well as music for 5 minutes and through the injection
  Interventions: Behavioral: Aromatherapy; Behavioral: Music
- control group (Other): children in this group will receive IANB injections with behavioral management techniques l
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Aromatherapy — Aroma therapy will apply before 5 minutes and during IANB injection in children, aromatherapy will apply through a nasal mask similar to one that uses when applying nitrous oxide after putting a 3d printed perforated box on the mask's circular halo on its surface, in this box cotton bolls impregnated with 3 drops of a 15% lavender-neroli oils blend are placed and then the child will smell the scent of aromatic oil blend from the box's perforated bottom surface which faces child's nose
  Arms: aromatherapy group; combination group music and aromatherapy
Behavioral: Music — Music will be played from a speaker in the treatment environment and will start 5 minutes before anesthesia and will be played through the whole anesthesia process, the music used will be chosen by the child from his favourite cartoon
  Arms: combination group music and aromatherapy; music group
Behavioral: Control — using a tell-show-do approach and children will put on a nasal mask without the box that contains an aromatic oil blend for the placebo effect
  Other Names: Placebo
  Arms: control group

SUMMARY:
The study sample will be divided randomly into 4 groups, each group will contain 27 children who need treatment in mandibular teeth and require anesthesia with inferior alveolar nerve block which is considered a painful procedure.

In the aromatherapy group, 3 drops of lavender-Neroli will be applied to cotton balls, which will be placed in a box designed with 3D printing to be placed on the nasal mask that is similar to the one used when administering nitrous oxide, so that the child inhales the aroma of the essential oil through the nasal mask. The mask is applied 5 minutes before administering local anesthesia in order to allow the child to inhale the oil aroma prior to and during local anesthesia.

In the music group, the music will be played from the recorder prior to local anesthesia and during it, music will be chosen by the child from the cartoon movies/tv shows they watch so that it is from his environment and familiar to them.

In The third group, both music and aromatherapy will drive the anesthesia process.

In The control groups, the child will put on the same nasal mask without an aromatherapy box to obtain a placebo effect and then receive the anesthesia.

DETAILED DESCRIPTION:
The sample of this study were children attending the department of pediatric dentistry faculty of dentistry, Damascus university, who need treatment in the mandibular teeth with an IANB injection After taking informed consent from the parent, the children were divided into 4 groups: aromatherapy intervention, music intervention, both aroma, and music intervention, and control groups

In the aromatherapy group:

firstly the essential oils were obtained from Biocham Natural Extracts co, Damascus, Syria(100%pure lavender (L.angustifolia), 100% pure Neroli (C. aranium)) and the main components of the oils were determined by gas chromatography, which was found to be 47% linalool acetate in lavender oil, and 37% linalool 9% limonene in Neroli oil Then A 15% lavender-Neroli oil was prepared by blending 2.3 ml lavender oil with 0.9 ml Neroli oil and diluting with grape seed oil to 20 ml which was done in the department of pharmacognosy, Faculty of pharmacy Damascus university In the dental treatment, A child will be allowed to inhale the aromatic scent of the oil blend through a cylindrical box which is 3D printed and contains cavities inside it and perforated from its upper and lower surface. It will be applied to the circular hole of the mask which is similar to the one that uses when supplying nitrous oxide. so that this box allows for safer aromatherapy, as it can be removed in the event of any allergy symptoms appearing on the child and provide him oxygen through the mask.

3 drops of 15%lavender-Neroli blend were poured on cotton balls and then put on the aroma box, the box then was placed on the mask which was applied to the child's nose, so that the child inhales the scent of the aromatic blend through the holes in the bottom of the box, which faces the child's nose.

The children were asked to inhale the aromatic oils blend 5 minutes before intervention and during needle insertion when administrating IANB injection.

In the music group:

The child asks to choose a song from their cartoons and program to make it familiar to them and desirable and then listen to it through a recorder So that the music is heard as a background in the environment surrounding the work to avoid isolating the child from his environment and the ability to continue audio communication between the doctor and the child.

The songs will play 5 minutes before and during needle administrating. In the combination group: aromatherapy and music were used above In the control group: the children who received IANB injection-s will be treated with child behavior management like tell-show-do and the nitrous oxide nasal mask was used without the box which was used to carry inside it the scent of the aromatic oils blend to obtain a placebo effect.

The child's anxiety level would be assessed through FLACC, Facial image scale, heart rate, systolic, Diastolic blood pressure, and respiratory saturation before and after injection.

The IANB injection was performed using a 27-gauge needle and a local anesthetic of 2% lidocaine with 1:100,000 epinephrine by one researcher.

ELIGIBILITY:
Inclusion Criteria:

* 1) 6-11 age children
* 2)children category 2,3 on Frankle behavior rating scale,
* 3) need treatment in mandibular molars to need anesthesia with IANB injection

Exclusion Criteria:

* 1) children with the mental or systematic disease
* 2) with a history of allergy, asthma, or have influenza
* 3)having a hearing problem or refusing to listen to music

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Self report anxiety assessment | directly 1second after anesthesia administration
  5 faces rang from very happy to very sad, one point is given to the most postive face and 5 point gives to the most negative face
Observation pain assessment | 5 second from starting the anesthesia
  Face, Legs, Activity, Cry, Consolability(FLACC), it has five categories of behavior to assess pain, namely , facial expression, leg movement, activity, cry, and Consolability, the score of each category are between 0and 2, the total score can rang from 0 to 10, defined as mild(1-3), moderate (4-6), and severe (7-10). for each patient, FLACC would be assess through video recorded during administration the IANB injection and then were evaluated by an external evaluator to determine the children behavior score according to this scale

SECONDARY OUTCOMES:
change in diastolic blood pressure | 5 minutes before anesthesia/20 second after anesthesia
  digital blood pressure monitor will be placed in the child's left elbow and the difference between the reading 5 minutes before anesthesia and after 20 sec from it
change in systolic blood pressure | 5 minutes before anesthesia/20 second after anesthesia
  digital blood pressure monitor will be placed in the child's left elbow and the difference between the reading 5 minutes before anesthesia and after 20 sec from it
change in pulse rate | 5 minutes before anesthesia/20second after anesthesia
  an oximeter will be placed on the finger of the left hand and the difference between the pulse reading 5 minutes before anesthesia and 20 sec after it
change in O2 saturation | 5 minutes before anesthesia/20 second after anesthesia
  an oximeter will be placed on the finger of the left hand and the difference between the saturation reading 5 minutes before anesthesia and 20 sec after it

CONTACTS AND LOCATIONS:
Overall Officials: Chaza Kouchaji, Professor, Study Director — Supervisal; Rasha Al-khatib, professor, Study Director — Co- supervisal
Locations (1):
- College of Dentistry, Damascus, Al-Mazzeh Saint, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ainscough SL, Windsor L, Tahmassebi JF. A review of the effect of music on dental anxiety in children. Eur Arch Paediatr Dent. 2019 Feb;20(1):23-26. doi: 10.1007/s40368-018-0380-6. Epub 2018 Oct 29. PMID 30374854
- [Background] Agatonovic-Kustrin S, Kustrin E, Gegechkori V, Morton DW. Anxiolytic Terpenoids and Aromatherapy for Anxiety and Depression. Adv Exp Med Biol. 2020;1260:283-296. doi: 10.1007/978-3-030-42667-5_11. PMID 32304038
- [Background] Arslan I, Aydinoglu S, Karan NB. Can lavender oil inhalation help to overcome dental anxiety and pain in children? A randomized clinical trial. Eur J Pediatr. 2020 Jun;179(6):985-992. doi: 10.1007/s00431-020-03595-7. Epub 2020 Feb 6. PMID 32030454
- [Background] Bradt J, Teague A. Music interventions for dental anxiety. Oral Dis. 2018 Apr;24(3):300-306. doi: 10.1111/odi.12615. Epub 2017 Jan 5. PMID 27886431
- [Background] Grisolia BM, Dos Santos APP, Dhyppolito IM, Buchanan H, Hill K, Oliveira BH. Prevalence of dental anxiety in children and adolescents globally: A systematic review with meta-analyses. Int J Paediatr Dent. 2021 Mar;31(2):168-183. doi: 10.1111/ipd.12712. Epub 2020 Sep 9. PMID 33245591
- [Background] Morgan AG, Rodd HD, Porritt JM, Baker SR, Creswell C, Newton T, Williams C, Marshman Z. Children's experiences of dental anxiety. Int J Paediatr Dent. 2017 Mar;27(2):87-97. doi: 10.1111/ipd.12238. Epub 2016 Jul 4. PMID 27376925
- [Background] Zhang N, Yao L. Anxiolytic Effect of Essential Oils and Their Constituents: A Review. J Agric Food Chem. 2019 Dec 18;67(50):13790-13808. doi: 10.1021/acs.jafc.9b00433. Epub 2019 Jun 13. PMID 31148444
- [Background] Suntar I, Khan H, Patel S, Celano R, Rastrelli L. An Overview on Citrus aurantium L.: Its Functions as Food Ingredient and Therapeutic Agent. Oxid Med Cell Longev. 2018 May 2;2018:7864269. doi: 10.1155/2018/7864269. eCollection 2018. PMID 29854097
- [Background] Ota M, Sato N, Sone D, Ogura J, Kunugi H. (-)-Linalool influence on the cerebral blood flow in healthy male volunteers revealed by three-dimensional pseudo-continuous arterial spin labeling. Indian J Psychiatry. 2017 Apr-Jun;59(2):225-227. doi: 10.4103/psychiatry.IndianJPsychiatry_323_16. PMID 28827872